CLINICAL TRIAL: NCT00519207
Title: Evaluation of Topical Liposomal Lidocaine and Oral Sucrose for Treatment of Pain in Newborn Infants Undergoing Venipuncture: A Randomized Controlled Trial
Brief Title: Evaluation of Topical Liposomal Lidocaine and Oral Sucrose for Treatment of Pain in Newborns Undergoing Venipuncture
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Anna Taddio/Principal Investigator, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1000010747
Record Dates: First submitted 2007-08-20; First posted 2007-08-22 (Estimated); Last update posted 2011-07-19 (Estimated); Status verified 2011-07

CONDITIONS: Pain
Keywords: pediatrics; pain; infants; newborn screening; venipuncture; lidocaine; sucrose
MeSH Terms: conditions — Pain | interventions — Lidocaine; Sucrose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): This group will receive lidocaine and sucrose placebo (water).
  Interventions: Drug: Lidocaine
- 2 (Active Comparator): This group will receive lidocaine placebo and sucrose.
  Interventions: Drug: 24% Sucrose Solution
- 3 (Active Comparator): This group will receive lidocaine and sucrose.
  Interventions: Drug: Lidocaine; Drug: 24% Sucrose Solution

INTERVENTIONS:
Drug: Lidocaine — 1g of liposomal lidocaine will be administered 30-40 minutes prior to venipuncture and occluded by a dressing.
  Other Names: Maxilene 4
  Arms: 1; 3
Drug: 24% Sucrose Solution — 2ml of 24% sucrose will be administered 2 minutes prior to venipuncture
  Other Names: TootSweet
  Arms: 2; 3

SUMMARY:
The objective of this study is to determine the relative efficacy of sucrose, liposomal lidocaine, and sucrose plus liposomal lidocaine, on reducing pain during venipuncture in newborn infants.

DETAILED DESCRIPTION:
Despite the fact that modern medical practice is greatly advanced, pain is inflicted on all Canadian newborn infants in the first days and months of life from blood tests, injections and cannulations designed to prevent, diagnose or manage medical conditions. Procedural pain in newborn infants is a significant burden to infants, their parents, healthcare workers, and society at large.

This study proposes a large randomized controlled trial to determine the optimal analgesic regimen for procedural pain using methods that can be easily implemented in clinical practice. We will study liposomal lidocaine cream and sucrose oral liquid, used alone, or together, to manage procedural pain. Liposomal lidocaine is a relatively new anaesthetic formulation ideally suited for young infants due to the established role of lidocaine in neonatal clinical medicine. Sucrose (sugar water) reduces pain responses and is promoted in consensus guidelines developed by pain experts. However, it is perceived by many front-line clinicians to be simply a comforting agent rather than a true analgesic. Studying liposomal lidocaine and sucrose together is important since the combination may prove superior to either agent alone, and may even prevent or abolish pain from clinical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Healthy newborn infants
* ≥ 37 weeks gestational age.

Exclusion Criteria:

* neonatal intensive care unit (NICU) admission
* asphyxia, seizures
* major birth defect (heart, brain, genetic syndrome)
* circumcised during study
* receiving analgesia/sedatives.

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 330 (Actual)
Dates: Start 2007-08; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Infant pain during venipuncture as assessed by facial grimacing response. | During venipuncture

SECONDARY OUTCOMES:
Visual Analog Scale scores | During venipuncture
Cry duration | During venipuncture
Heart rate | During venipuncture
Number of attempts until procedure completion | From first needle poke to completion
Endomorphins-1,-2 levels | Before and 10 minutes after sucrose/sucrose placebo administration
Procedure duration | From first needle poke to completion
Lidocaine levels | 5-15 minutes after the study cream is removed

CONTACTS AND LOCATIONS:
Overall Officials: Anna Taddio, PhD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (2):
- Canada (2):
  - Mount Sinai Hospital, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario